CLINICAL TRIAL: NCT02536547
Title: Diagnostic Value of Pulmonary Ultrasound in the Diagnosis of Ventilator-associated Pneumoniae
Acronym: PAVM
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Collaborators: Istituto Nazionale di Ricovero e Cura per Anziani (Other)
Responsible Party: Sponsor
Other Study IDs: 2013-A01818-37
Record Dates: First submitted 2015-08-21; First posted 2015-09-01 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Ventilator-associated Pneumonia; Sepsis
Keywords: Clinical pulmonary infection score; sepsis; lung ultrasound; ventilator-associated pneumonia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — biochemistry : procalcitonin, leukocytes, neutrophils
  microbiology : bronchoalveolar lavage and tracheal aspiration
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients with suspected VAP: All patients with suspected VAP will be included in the study (new or extension of a radiological image in a patient in mechanical ventilation for at least 48 hours associated with at least two of the following:criteria :
  fever ≥38.5 ° C or <36, 5 ° C leukocytosis> 10 * 103 / ml or leukopenia <4 * 103 / ml secretions purulent tracheal reduction in PaO2 / FiO2 <300 or PaO 2 <60 mmHg
  Interventions: Device: VAP

INTERVENTIONS:
Device: VAP — all patients with suspected VAP : biochemestry microbiology lung ultrasound

SUMMARY:
This study evaluates the respective values and combined CPIS (Clinical Pulmonary Infection Score), bronchoalveolar lavage (BAL), tracheal aspiration and pulmonary ultrasonography (LUS - Lung Ultrasound) for early diagnosis of ventilator- associated pneumonia (VAP).

DETAILED DESCRIPTION:
Diagnosis and monitoring iconographic lung infection is essentially limited to chest radiography. But this one to bed is a source of information generally unreliable routine.

Lung ultrasound is now an additional technique for confirmation of diagnosis and followed by community acquired pneumonia and monitoring of ventilator-associated pneumonia. The specific pathophysiology of VAP makes particularly efficient lung ultrasound in the diagnosis and monitoring of these attacks. The patient mechanically ventilated, the colonization of the airways is responsible for a continuous seeding of the tracheobronchial tree. As the lesions are scattered throughout the lung parenchyma and are centered on a bronchiole; although there is a predominance of households in the areas most dependent lung. VAP is therefore characterized by inflammatory tissue expansion to the periphery, predominant at the lower lobes and partnering with a ventilation loss varies with the severity of the pneumonia.

Thus, it can be found at an early stage some cells infected around a bronchiole in contact with infected acini normally ventilated. At an advanced stage, this extension to the whole parenchyma results in the widespread presence of small outbreaks in pleural. They are easily and specifically detected by ultrasound in the form of vertical artifacts irregular spacing (irregular Lines B) or small pictures (<0.5 cm) rounded HYPOECHOIC (jucta pleural consolidation) for reliable diagnosis of VAP. The success of an antibiotic is detected by the disappearance of B lines and pleural jucta consolidations. The failure of antibiotic therapy by the appearance of new jucta pleural consolidations which may merge giving lobar consolidation. Community-acquired pneumonia is characterized by the spread of infection in a home adjacent pulmonary segments by providing a systematized typical lobar reached. The diagnosis and monitoring of community-acquired pneumonia is mainly based on monitoring the number and size of household lobar consolidation which is not sufficient for pneumonia Ventilator. This latest study shows that the intensity ultrasound signs is proportional to the extension of outbreaks (lobar consolidations homes and mini homes jucta pleural consolidation). Moreover unlike biological biomarkers such as procalcitonin, it does not reflect the intensity of inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Patients in mechanical ventilation for at least 48 hours
* and new or extension of a radiological image

with at least two of the following clinical criteria:

* Body temperature ≥ 38.5 ° C or <36 ° C
* Leukocytes> 10 * 103 / ml or <4 * 103 / ml or> 10% immature cells (in the absence of other known causes).
* hypoxemia with PaO 2 <60 mmHg or a P / F <300
* secretions purulent tracheal

Exclusion Criteria:

* Patient with known pneumonia
* Patient under 18 years
* Mechanical ventilation <48h
* contraindication of pulmonary endoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with suspected VAP will be included in the study (new or extension of a radiological image in a patient in mechanical ventilation for at least 48 hours associated with at least two of the following criteria : fever ≥38.5 ° C or <36, 5 ° C, leukocytosis> 10 * 103 / ml or leukopenia <4 * 103 / ml; secretions purulent tracheal; reduction in PaO2 / (FiO2) <300 or PaO2 <60 mmHg)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Sensitivity, specificity and diagnostic accuracy of lung ultrasound (in pleural consolidation homes and irregular lines B, basal consolidation) only and associated with the CPIS (clinical pulmonary infection score) | 48h after mecanic ventilation

SECONDARY OUTCOMES:
Frequency of specific sonographic signs (irregular B lines, pleural consolidation in household) during the VAP | 48h after mecanic ventilation
Diagnostic approach integrating CPIS (Clinical Pulmonary Infection Score), tracheal aspiration and lung ultrasound (LUS - Lung Ultrasound) for the early diagnosis of VAP | 48h after mecanic ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Bélaïd BOUHEMAD, Dr, Principal Investigator — Fondation Hôpital Saint-Joseph